CLINICAL TRIAL: NCT03031392
Title: Sensitivity and Specificity of Peri-Implantitis-Related Parameters: A Case-Control Study
Brief Title: Sensitivity and Specificity of Peri-Implantitis-Related Parameters
Status: Completed | Type: Observational
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Sponsor
Other Study IDs: 18002909/3
Record Dates: First submitted 2017-01-20; First posted 2017-01-25 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-01

CONDITIONS: Sensitivity; Peri-implant Mucositis; Peri-Implantational Loss; Peri-Implantitis
MeSH Terms: conditions — Hypersensitivity; Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peri-implantitis: Individuals with implants ≥2mm of radiographic bone loss
  Interventions: Diagnostic Test: Sensitivity test
- non-peri-implantitis patients: Individuals with implants <2mm of radiographic bone loss
  Interventions: Diagnostic Test: Sensitivity test

INTERVENTIONS:
Diagnostic Test: Sensitivity test — Routine clinical and radiographic examination

SUMMARY:
Bleeding on probing demonstrated to have high specificity with certain level of sensitivity to detect periodontal disease. Again, understanding the weak hemidesmosome attachment to the implant surface is imperative to discern on the probe penetration extent and subsequent bleeding. In the presence of inflammation, bleeding should be present indicating high sensitivity when probing deeper sites; nevertheless the lack thereof in healthy condition does not seem to translate high specificity. In this sense, it is noteworthy to mention that the mucogingival shift after implant placement often decreases the presence of keratinized mucosa, triggering a greater inflammatory condition on the peri-implant tissues. Thereupon, bleeding on probing, although might reliably indicate presence of disease, it does not seem to be a suitable diagnostic parameter. On the other side, suppuration characterizes the necrosis of peri-implant tissues, being rich in polymorphonuclear cells and as such, a sensitive indicator of bone turnover. In this sense, it must be noted that, if detected in early stages where bone resorption has not occurred yet, it might be a consequence of a foreign body reaction (i.e., residual cement or floss).

Therefore, in the diagnosis of peri-implantitis, radiographic examination must be always incorporated to the clinical assessment as the 'gold standard'. Hence, the aim of this case-control study was to assess the diagnostic accuracy of peri-implantitis-related clinical parameters compared to otherwise healthy dental implants.

DETAILED DESCRIPTION:
All subjects enrolled had to be consecutively evaluated in a routine peri-implant maintenance t with dental implants for fixed prosthesis rehabilitation with a minimum period of 12 months after final prosthesis delivery. Patients were contacted and informed to participate in a cross-sectional assessment to identify the presence of peri-implant diseases. Eligible implants had to be in an ideal prosthetically driven position, otherwise they were excluded from the analysis. Moreover, implants that could not be accurately recorded the probing depth due to inadequate prosthesis design were further excluded. Baseline periapical x-ray at time of prosthesis delivery was retrospective assessed to exclude implants with early peri-implant bone loss before function. A detailed description of risk factors and indicators of peri-implant disease were explained at the same stage. Additionally, patients were thoroughly instructed on plaque control home care strategies including but not limited to interdental brushes with nylon-coated core wire, soft toothbrushes (manual and power) and floss with stiffened end to clean under multiple units fixed-prosthesis. Moreover, treated patients were encouraged to routinely enroll in a peri-implant maintenance therapy program.

The present case-control study will be conducted in accordance with the Helsinki declaration of human studies and received approval from the ethics committee from the University of Extremadura (Badajoz, Spain). An informed written consent was signed from each subject enrolled in the present study.

ELIGIBILITY:
Inclusion Criteria:

* patients within the age range of 18 to 80,
* non- or light smokers (<10cigarettes/day),
* no presence of infectious diseases at the time of implant placement or during the maintenance program,
* no presence of serious disease or condition known to alter bone metabolism,
* partial edentulous patients with stable periodontal condition with or without history of chronic periodontitis.

Exclusion Criteria:

* pregnancy,
* history of heavy smoking,
* uncontrolled medical conditions such as diabetes mellitus,
* not adequate implant position (i.e., prosthetically driven),
* not properly restored impeding accurate probing depth recording
* lack of keratinized mucosa

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be either approached during their biannual peri-implant maintenance recall appointment or contacted and asked to participate in a free clinical and radiographic examination to identify the possible presence of peri-implant pathology.
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity to detect peri-implantitis | 1 year
  Capability to diagnose disease
Specificity to detect peri-implantitis | 1 year
  Capability to diagnose health

CONTACTS AND LOCATIONS:
Overall Officials: Florencio Monje Gil, Study Director — Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain
Locations (1):
- Centro de Implantologia Cirugia Oral y Maxiofacial, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No